CLINICAL TRIAL: NCT00845312
Title: Prognostic Features for Mortality in Adult Pneumonia Patients at the Age of Sixty and Beneath.
Brief Title: Prognostic Features for Mortality in Young Adults With Pneumonia
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Eyal Braun M.D., Internal Medicine "B", Rambam Health Care Campus
Other Study IDs: CTIL
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2009-02

CONDITIONS: Pneumonia
Keywords: Age; Mortality
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Complicated hospitalization: Patients 60 years old or younger, who were diagnosed with community acquired pneumonia (CAP) between March 1, 2005 and December 31, 2008 were retrospectively analyzed for risk factors for severe morbidity or mortality.
  was defined as at least one of the following parameters: hospitalization longer than ten days, admission to intensive care unit and in- hospital mortality. Otherwise, the hospitalization was defined uncomplicated .The Rambam hospital Institutional Review Board approved the study.

SUMMARY:
Pneumonia is a major cause of mortality and morbidity. A large body of evidence concerning the mortality risk factors in elderly patients with pneumonia has been reported; however, less is known about causes of mortality in patients of sixty and less. We noted a relatively substantial rate of short term mortality in this group of patients that were admitted to our institution. Therefore, we aimed to estimate the mortality rate and to identify risk factors for mortality among patients of sixty years old and less that were admitted with community acquired pneumonia.

DETAILED DESCRIPTION:
Community acquired pneumonia (CAP) is a major cause of morbidity and mortality. While there is much data about risk factors for severe outcome in the general population, there is less focus on younger group of patients. Therefore, we aimed to detect simple prognostic factors for severe morbidity and mortality in young patients with CAP.

Patients 60 years old or younger, who were diagnosed with CAP (defined as Pneumonia identified 48 hours or less from hospitalization) between March 1, 2005 and December 31, 2008 were retrospectively analyzed for risk factors for severe morbidity or mortality.

Complicated hospitalization was defined as at least one of the following parameters: hospitalization longer than ten days, admission to intensive care unit and in- hospital mortality. Otherwise, the hospitalization was defined uncomplicated

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of community acquired pneumonia Age between 18-60

Exclusion Criteria:

Age less than 18 and more than 60 Transfer from another hospital Hospitalization for any cause other than CAP during the 30 days prior to admission Hospital acquired pneumonia Partial antibiotic treatment before admission.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that were admitted with community acquired pneumonia to Rambam Medical Center between the dates January 1, 2004 until December 31, 2008
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaher S Azzam, MD, Study Chair — Head Of Internal Medicine "B"; Eyal Braun, MD, Principal Investigator — Deputy Head of Internal Medicine "B"
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Braun E, Domany E, Kenig Y, Mazor Y, Makhoul BF, Azzam ZS. Elevated red cell distribution width predicts poor outcome in young patients with community acquired pneumonia. Crit Care. 2011 Aug 11;15(4):R194. doi: 10.1186/cc10355. PMID 21835005